CLINICAL TRIAL: NCT02431078
Title: The Expression of Zinc Finger E-Box Binding Homeobox 1 (ZEB1) in Circulating Tumor Cells(CTCs) Associated With Metastasis and Recurrence for Gastric Cancer
Brief Title: The Expression of ZEB1 in CTCs Associated With Metastasis and Recurrence for Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: wei bo (Other)
Responsible Party: Sponsor-Investigator, wei bo, Vice Director of the general surgery department, Chinese PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: experiment20152018
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-04

CONDITIONS: Stomach Neoplasms
Keywords: CTCs; ZEB1; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating Tumor Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ZEB1 high-expression group: Participants with ZEB1 high-expression(ZEB1 expression values>the ZEB1 cut-off point) in CTCs for gastric cancer will be assigned to this group.The ZEB1 cut-off point was set at the top quartile.Routine comprehensive treatment will be performed.
  Interventions: Procedure: Routine comprehensive treatment
- ZEB1 low-expression group: Participants with ZEB1 low-expression(ZEB1 expression values<the ZEB1 cut-off point) in CTCs for gastric cancer will be assigned to this group.The ZEB1 cut-off point was set at the top quartile.Routine comprehensive treatment will be performed.
  Interventions: Procedure: Routine comprehensive treatment

INTERVENTIONS:
Procedure: Routine comprehensive treatment — Radical gastrectomy for gastric cancer and postoperative adjuvant chemotherapy

SUMMARY:
The aim of this study was to investigate the expression of ZEB1 in CTCs for gastric cancer, its correlation with the clinicopathology of gastric cancer, and the role of ZEB1 in invasion and metastasis in gastric cancer.

DETAILED DESCRIPTION:
Invasion and metastasis of tumors and postoperative recurrence are the main causes of death in patients with gastric cancer and are also the key factors affecting the clinical treatment and prognosis.

In this study, the investigators will detect the expression of ZEB1 in different types of CTCs(epithelial,mesenchymal and mixed phenotype) for gastric cancer by CanPatrolTM2 detection technology.Our investigation of the relationship between ZEB1 and the occurrence and development as well as the invasion and metastasis of gastric cancer is expected to provide data for the prognosis and targeted therapy of gastric cancer.

Approximate 100 consecutive patients with gastric cancer and CTCs(+) will be enrolled in this study.Detection of ZEB1 expression in CTCs at baseline will show the relationship between ZEB1 and clinicopathological variables. Postoperative follow-up of ZEB1 expression in CTCs will be performed every three months in the first year and every six months in the following two years. The results may indicate the role of ZEB1 in CTCs about invasion and metastasis for gastric cancer .The aim of this study is to clarify the clinical significance of ZEB1 expression in CTCs for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven gastric cancer and CTCs(+).
2. Age:older than 18 years old,younger than 80 years old.
3. cT1-4a(surgically resectable tumor),N0-3,M0 at preoperative evaluation according to the American Joint Committee on Cancer(AJCC) Cancer Staging Manual Seventh Edition.
4. No obvious surgical contraindications.
5. American Society of Anesthesiology (ASA) score class I, II, or III.
6. Written informed consent.

Exclusion Criteria:

1. Severe mental disorder.
2. Pregnancy.
3. History of previous gastrectomy,endoscopic mucosal resection or endoscopic submucosal dissection.
4. History of unstable angina or myocardial infarction within past six months.
5. History of previous neoadjuvant chemotherapy or radiotherapy.
6. History of other malignant disease within past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximate 150 consecutive patients with gastric cancer and CTCS(+) will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
three-year disease free survival rate | Up to 3 years post-operative

SECONDARY OUTCOMES:
three-year overall survival rate | Up to 3 years post-operative
metastasis and recurrence rate | Up to 3 years post-operative
baseline detection of ZEB1 expression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wei bo, MD, Study Chair — Vice director of the general surgery department, Chinese PLA General Hospital

REFERENCES:
- [Background] Barriere G, Fici P, Gallerani G, Fabbri F, Zoli W, Rigaud M. Circulating tumor cells and epithelial, mesenchymal and stemness markers: characterization of cell subpopulations. Ann Transl Med. 2014 Nov;2(11):109. doi: 10.3978/j.issn.2305-5839.2014.10.04. PMID 25489583
- [Background] Toss A, Mu Z, Fernandez S, Cristofanilli M. CTC enumeration and characterization: moving toward personalized medicine. Ann Transl Med. 2014 Nov;2(11):108. doi: 10.3978/j.issn.2305-5839.2014.09.06. PMID 25489582
- [Background] Okugawa Y, Toiyama Y, Tanaka K, Matsusita K, Fujikawa H, Saigusa S, Ohi M, Inoue Y, Mohri Y, Uchida K, Kusunoki M. Clinical significance of Zinc finger E-box Binding homeobox 1 (ZEB1) in human gastric cancer. J Surg Oncol. 2012 Sep 1;106(3):280-5. doi: 10.1002/jso.22142. Epub 2011 Nov 17. PMID 22095522
- [Background] Yabusaki N, Yamada S, Murai T, Kanda M, Kobayashi D, Tanaka C, Fujii T, Nakayama G, Sugimoto H, Koike M, Nomoto S, Fujiwara M, Kodera Y. Clinical significance of zinc-finger E-box binding homeobox 1 mRNA levels in peritoneal washing for gastric cancer. Mol Clin Oncol. 2015 Mar;3(2):435-441. doi: 10.3892/mco.2014.462. Epub 2014 Nov 20. PMID 25798282
- [Background] Jia B, Liu H, Kong Q, Li B. Overexpression of ZEB1 associated with metastasis and invasion in patients with gastric carcinoma. Mol Cell Biochem. 2012 Jul;366(1-2):223-9. doi: 10.1007/s11010-012-1299-6. Epub 2012 Mar 31. PMID 22466758
- [Background] Yang X, Wang Q, Dai W, Zhang J, Chen X. Overexpression of zinc finger E-box binding homeobox factor 1 promotes tumor invasiveness and confers unfavorable prognosis in esophageal squamous cell carcinoma. Tumour Biol. 2014 Dec;35(12):11977-84. doi: 10.1007/s13277-014-2494-8. Epub 2014 Aug 21. PMID 25142232
- [Background] Beije N, Jager A, Sleijfer S. Circulating tumor cell enumeration by the CellSearch system: the clinician's guide to breast cancer treatment? Cancer Treat Rev. 2015 Feb;41(2):144-50. doi: 10.1016/j.ctrv.2014.12.008. Epub 2014 Dec 23. PMID 25542852
- [Background] Graham TR, Zhau HE, Odero-Marah VA, Osunkoya AO, Kimbro KS, Tighiouart M, Liu T, Simons JW, O'Regan RM. Insulin-like growth factor-I-dependent up-regulation of ZEB1 drives epithelial-to-mesenchymal transition in human prostate cancer cells. Cancer Res. 2008 Apr 1;68(7):2479-88. doi: 10.1158/0008-5472.CAN-07-2559. PMID 18381457